CLINICAL TRIAL: NCT02805192
Title: Validation of a Smart Phone App to Non-invasively Measure the Size of Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Zurich (Other)
Responsible Party: Principal Investigator, Philipp Stein, Dr. med. Philipp Stein, University of Zurich
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: KEK 2016-271, 94-2015
Record Dates: First submitted 2016-06-10; First posted 2016-06-17 (Estimated); Last update posted 2017-05-03 (Actual); Status verified 2017-05

CONDITIONS: Growth and Development
Keywords: Emergency Department; Estimation of age and weight; Size measurement
MeSH Terms: conditions — Emergencies; Body Weight

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- one Arm: size measurement by Smart phone App (Other)
  Interventions: Device: Size Measurement by a Smart phone App

INTERVENTIONS:
Device: Size Measurement by a Smart phone App

SUMMARY:
Smart phones are omnipresent. Apps exist to calculate size of medical equipment and doses of medication if a valid weight or age is entered. During emergency situations, these values are often unknown. An App has been developed to measure the size of a child noninvasively. This App is now to be validated in clinical practice. App measured size is calculated and compared to the real size of a child. Via known percentiles of age/weight of the child is calculated upon the App measured size. This value is compared to the mother's, physician's and nurses estimation of the size and weight.

Depending on the size multiple algorithms exist to estimate weight, age and medical values. ("Kindersicher ®", "Notfalllineal ®" and "Broselow Tape ®"). These estimations by the calculations will also be compared to actual weight and age.

Children from 0-12 years of age are included in the emergency Department of the Children's Hospital of the University of Zurich after informed consent obtained by the parents. No therapy decisions from these calculations will be made. The therapy is independent of this study.

ELIGIBILITY:
Inclusion Criteria:

* male and female patients 0-12 years of age (45 per age group)
* obtained informed consent
* admitted to the emergency department of the Children's Hospital of the University of Zurich

Exclusion Criteria:

* physically or mentally unable for measurement
* denial of informed consent

Max Age: 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 627 (Actual)
Dates: Start 2016-01-30; Primary Completion 2016-06-30 (Actual); Study Completion 2016-06-30 (Actual)

PRIMARY OUTCOMES:
Comparison of the size measured by the smart phone app with the child's size. | immediate, no follow up

SECONDARY OUTCOMES:
Comparison of the estimations calculated upon the smart phone measured size (via known percentiles) with the real age and weight. | immediate, no follow up
Comparison of estimations by "Kindersicher ®", "Notfalllineal ®" and "Broselow Tape ®" with real age and weight. | immediate, no follow up
Comparison of estimations by parents, physicians and nurses with the actual size and weight. | immediate, no follow up

CONTACTS AND LOCATIONS:
Overall Officials: Donat R Spahn, M.D., F.R.C.A., Study Chair — University and Universtity Hospital Zurich
Locations (1):
- Universtity Hospital Zurich, Zurich, Switzerland

REFERENCES:
- [Derived] Wetzel O, Schmidt AR, Seiler M, Scaramuzza D, Seifert B, Spahn DR, Stein P. A smartphone application to determine body length for body weight estimation in children: a prospective clinical trial. J Clin Monit Comput. 2018 Jun;32(3):571-578. doi: 10.1007/s10877-017-0041-z. Epub 2017 Jun 28. PMID 28660564